CLINICAL TRIAL: NCT01193959
Title: Retrospective Study of Molecular Predictors of Sensitivity and Resistance to Pemetrexed in Advanced Non-Small Cell Lung Cancer
Brief Title: Pemetrexed in Advanced Non-small Cell Lung Cancer
Status: Completed | Type: Observational
Sponsor: Armando Santoro, MD (Other)
Responsible Party: Sponsor-Investigator, Armando Santoro, MD, MD, Istituto Clinico Humanitas
Organization: Istituto Clinico Humanitas (Other)
Other Study IDs: ONC/OSS-02/2010
Record Dates: First submitted 2010-08-26; First posted 2010-09-02 (Estimated); Last update posted 2022-09-10 (Actual); Status verified 2022-09

CONDITIONS: Non-small Cell Lung Cancer (NSCLC)
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Present study is aimed at investigating potential molecular predictors of sensitivity or resistance to single-agent pemetrexed in the ≥ second line setting in a large cohort of advanced non-small cell lung cancer (NSCLC) patients. The following biomarkers will be investigated with either immunohistochemistry, fluorescence in situ hybridization or genotyping: thymidylate synthase (TS), dihydrofolate reductase (DHFR), glycinamide ribonucleotide formyl transferase (GARFT), aminoimidazole carboxamide ribonucleotide formyltransferase (ATIC/AICARFT), epidermal growth factor receptor (EGFR), Kirsten rat sarcoma 2 viral oncogene homolog (KRAS), v-myc myelocytomatosis viral oncogene homolog (MYC) and phosphoinositide-3-kinase, catalytic, alpha polypeptide (PIK3CA).

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed diagnosis of advanced non-small cell lung cancer - Tumor tissue available at our institution
* Patients treated with single agent pemetrexed for metastatic disease
* Availability of full clinical data

Exclusion Criteria:

* Cytological diagnosis of advanced Non-small cell lung cancer
* Lack of tumor tissue at our institution
* Lack of full clinical data

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Non-small cell lung cancer patients treated with single agent pemetrexed
Sampling Method: Non-Probability Sample
Enrollment: 33 (Actual)
Dates: Start 2010-09; Primary Completion 2011-12 (Actual); Study Completion 2012-06 (Actual)

PRIMARY OUTCOMES:
Association of each biomarker with treatment outcome in terms of response rate, time to progression, overall survival. | one year

SECONDARY OUTCOMES:
Association of each biomarker with clinico-pathological features: histology, gender, age, smoking status, response to previous chemotherapy. | one year

CONTACTS AND LOCATIONS:
Overall Officials: Armando SANTORO, MD, Principal Investigator — Istituto Clinico Humanitas
Locations (1):
- Istituto Clinico Humanitas, Rozzano, Milano, Italy